CLINICAL TRIAL: NCT06517862
Title: Efficacy and Safety of Oral Zinc Sulphate and Ursodeoxycholic Acid as Adjuvants to Phototherapy in Management of Neonatal Non-Hemolytic Unconjugated Hyperbilirubinemia
Brief Title: Efficacy & Safety of Oral Adjuvants to Phototherapy in Neonatal Hyperbilirubinemia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Amira Adel Fouly (Other)
Collaborators: Egyptian Chinese University (Other); Ain Shams University (Other)
Responsible Party: Sponsor-Investigator, Amira Adel Fouly, principal investigator, Future University in Egypt
Organization: Future University in Egypt (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC-FPFUE-31/2023
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Neonatal Hyperbilirubinemia
Keywords: Neonatal hyperbilirubinemia; Phototherapy; exchange transfusion; Zinc sulfate; Ursodeoxycholic acid
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal | interventions — Zinc Sulfate; Ursodeoxycholic Acid

STUDY DESIGN:
Intervention Model Description: 8 arms (Full term Control, Full term Low Dose Zinc Sulphate, Full term High Dose Zinc Sulphate, Full term UDCA -- Preterm Control, Preterm Low Dose Zinc Sulphate, Preterm High Dose Zinc Sulphate, Preterm UDCA)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- preterm: control (No Intervention): phototherapy only
- preterm: low dose of oral zinc sulfate (Experimental): Neonates will receive oral Zn sulfate solution in low doses (10 mg/day) given as 5 mg twice daily.
  Interventions: Drug: Zinc sulfate
- preterm: high dose of oral zinc sulfate (Experimental): Neonates will receive oral Zn sulfate solution in a high dose (20 mg/day) given as 10 mg twice daily.
  Interventions: Drug: Zinc sulfate
- preterm: low dose of oral UDCA (Experimental): Neonates will receive oral UDCA solution at 10 mg/kg twice daily.
  Interventions: Drug: Ursodeoxycholic acid
- full-term: control (No Intervention): phototherapy only
- full-term: low dose of oral zinc sulfate (Experimental): Neonates will receive oral Zn sulfate solution in low doses (10 mg/day) given as 5 mg twice daily.
  Interventions: Drug: Zinc sulfate
- full-term: high dose of oral zinc sulfate (Experimental): Neonates will receive oral Zn sulfate solution in a high dose (20 mg/day) given as 10 mg twice daily.
  Interventions: Drug: Zinc sulfate
- full-term: low dose of oral UDCA (Experimental): Neonates will receive oral UDCA solution at 10 mg/kg twice daily.
  Interventions: Drug: Ursodeoxycholic acid

INTERVENTIONS:
Drug: Zinc sulfate — Neonates will receive oral Zn sulfate solution in either low doses (10 mg/day) or high doses (20 mg/day) given twice daily.
  Other Names: zinc origin
  Arms: full-term: high dose of oral zinc sulfate; full-term: low dose of oral zinc sulfate; preterm: high dose of oral zinc sulfate; preterm: low dose of oral zinc sulfate
Drug: Ursodeoxycholic acid — Neonates will receive oral UDCA solution at 10 mg/day given as 5 mg twice daily.
  Other Names: Livagoal
  Arms: full-term: low dose of oral UDCA; preterm: low dose of oral UDCA

SUMMARY:
Neonatal jaundice, or neonatal hyperbilirubinemia, is a common medical issue in the first two weeks of life, causing prolonged hospitalization and readmissions. It results from elevated total serum bilirubin (TSB) and is manifested as yellowish discoloration of the skin, sclera, and mucous membrane. Clinical jaundice appears in about 60% of term neonates and 80% of preterm infants within the first week of life. Pathologic hyperbilirubinemia occurs when bilirubin levels increase by more than 5 mg/dL/day or 0.2 mg/dL/hour, or when jaundice lasts longer than two to three weeks in full-term infants. In preterm infants, unconjugated hyperbilirubinemia is of particular concern due to their permeable blood-brain barrier and underdeveloped brain. Phototherapy is widely used to reduce or prevent the rise of serum unconjugated bilirubin levels and reduce the need for exchange transfusions. However, phototherapy has both immediate and long-term side effects, and it can only decrease accumulated UCB but does not prevent its accumulation. There is a growing potential to explore novel adjuvant treatments to increase bilirubin clearance, decrease phototherapy duration, and decrease exchange transfusion rate.

DETAILED DESCRIPTION:
Neonatal jaundice, or neonatal hyperbilirubinemia, is the most common medical issue in the first two weeks of life and is a frequent cause of prolonged hospitalization and readmission to the hospital after birth. It results from elevated total serum bilirubin (TSB) and is clinically manifested as yellowish discoloration of the skin, sclera, and mucous membrane. Increased enterohepatic circulation of indirect bilirubin is one of the elucidated mechanisms implicated in the pathophysiology of neonatal hyperbilirubinemia.

Clinical jaundice appears in about 60% of term neonates and 80% of preterms within the first week of life. In most cases, it is a mild, transient, and self-limiting condition that resolves spontaneously and is referred to as "physiological jaundice.". When bilirubin levels increase by more than 5 mg/dL/day or more than 0.2 mg/dL/hour, or when jaundice lasts longer than two to three weeks in full-term infants, pathologic hyperbilirubinemia is said to have occurred. In preterm infants, unconjugated hyperbilirubinemia is of particular concern, given that their blood-brain barrier is more permeable, and their underdeveloped brain is more susceptible to bilirubin-induced neurotoxicity.

Scavenging unconjugated plasma bilirubin can be done, conveniently, non-invasively, and effectively by phototherapy. Phototherapy is universally recognized as the mainstay for the treatment of neonatal jaundice and is widely used in neonatal units and postnatal wards. It is a safe and effective method for decreasing or preventing the rise of serum unconjugated bilirubin levels, and it reduces the need for exchange transfusions in neonates.

However, phototherapy has both immediate and long-term side effects, such as rash, bronze baby syndrome, and circadian rhythm modification. This is coupled with social side effects like parental concern because of the infant's increased hospitalization, broken mother-infant attachment, and high cost of care. Moreover, phototherapy can only decrease already accumulated UCB but does not prevent its accumulation. Exchange transfusion therapy, which is generally performed after the failure of phototherapy, may lead to severe complications, such as embolism, sepsis, necrotizing enterocolitis, or even death.

Consequently, there is a growing potential to explore novel adjuvant treatments that can help to increase bilirubin clearance, decrease phototherapy duration, and decrease exchange transfusion rate.

One of the methods used to treat indirect hyperbilirubinemia is to use a zinc solution. Studies have shown that chronic or acute use of zinc salts can reduce serum bilirubin levels by inhibiting the enterohepatic cycle of indirect bilirubin. Oral administration of zinc (Zn) sulfate increases bilirubin excretion and decreases its serum level.

Oral administration of Zn salts is possible in two dose ranges: low (10 mg/day) and high (11-20 mg/day). Given that some of the medication is absorbed in the proximal ileum, giving a high dose may be desirable. Zn salts are safe, and studies treating several children and newborns with diarrhea, measles, pneumonia, the common cold, and malaria have demonstrated the safety of oral Zn sulfate administration. Studies conducted on the effectiveness of Zn salts on serum indirect bilirubin levels in newborns have yielded different results, all calling for further research. Additionally, neonates with hyperbilirubinemia appear to have lower serum Zn levels than other well-term neonates.

The efficacy of ursodeoxycholic acid as an adjuvant to phototherapy has also been examined in a few studies. Ursodeoxycholic acid (UDCA), or ursodiol, is a bile acid commonly used to manage cholestatic liver disease. UDCA helps in improving endogenous bile secretion, reducing the reducing the displacement of more toxic components of endogenous bile acids, and reducing enterohepatic circulation. Because of its anti-apoptotic, anti-inflammatory, and antioxidant characteristics, UDCA also has hepatoprotective and neuroprotective effects.

Although UDCA is an off-label treatment in neonates, it is widely used in conjugated hyperbilirubinemia and liver disorders. UDCA has also been investigated for its possible role in indirect hyperbilirubinemia. It is thought to function by inhibiting the reabsorption of bilirubin from the intestines. UDCA is often tolerated well. In studies on healthy-term neonates, ill neonates, and neonates with G6PD deficiency, UDCA was reported to be useful in shortening the length of phototherapy.

ELIGIBILITY:
Inclusion Criteria:

* neonates with both genders
* neonates with gestational age ≥ 32 weeks
* neonates who can tolerate enteral feeding
* diagnosed with unconjugated non-hemolytic hyperbilirubinemia
* Phototherapy is required within the first week of life.

Exclusion Criteria:

* Neonates with seizures, hydrops fetalis, hypoxic-ischemic encephalopathy, or major congenital anomalies
* Neonates who have had an exchange transfusion within 24 hours
* neonates have evidence of hemolytic causes of jaundice (e.g., ABO and RH
* incompatibility, glucose 6-phosphate dehydrogenase deficiency)
* neonates who have reported hypersensitivity to zinc sulfate or ursodeoxycholic acid.

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
serum bilirubin level. | 10 days
  Assessing the effect of oral administration of zinc sulfate (at low and high doses) and ursodeoxycholic acid on serum bilirubin levels during the treatment of neonatal non-hemolytic unconjugated hyperbilirubinemia.
duration of phototherapy needed. | 10 days
  Assessing the effect of oral administration of zinc sulfate (at low and high doses) and ursodeoxycholic acid on the duration of phototherapy during the treatment of neonatal non-hemolytic unconjugated hyperbilirubinemia.

SECONDARY OUTCOMES:
monitoring adverse effects | 10 days
  assessing the possible side effects of both drugs
serum zinc level | 10 days
  evaluate the level of serum zinc before and after interventions.
length of NICU stay. | 10 days
  assess if the intervention will affect the duration of the NICU stay.

CONTACTS AND LOCATIONS:
Overall Officials: Ehab R. Bendas, professor, Study Director — Future University in Egypt; Yasmin A. Farid, Study Director — Ain Shams University; Dina K. Abou El Fadl, Lecturer, Study Director — Future University in Egypt; Sarah S. Hesham, Lecturer, Study Director — Egyptian Chinese University
Locations (1):
- Neonatal Intensive Care Unit (NICU) of Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No